CLINICAL TRIAL: NCT01407744
Title: Examination of the Multiple Genetic and Molecular Targets as Therapeutic Options for Patients With Ependymoma Treated by the Phase II Children's Oncology Group Study ACNS0121
Brief Title: Study of Tumor Samples From Patients With Ependymoma Treated on the Children's Oncology Group ACNS0121 Trial
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACNS11B1; NCI-2011-03801 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA098543 (NIH)
Record Dates: First submitted 2011-07-30; First posted 2011-08-02 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Infratentorial Ependymoma; Childhood Supratentorial Ependymoma; Newly Diagnosed Childhood Ependymoma

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archived tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative studies: Archived tumor tissue samples are analyzed by laboratory biomarker analysis for cellular density, mitotic count, tumor cell invasion, hTERT expression, telomere dysfunction, 1q gain, 9p deletion, and genetic mutations by IHC, Affymetrix MIP arrays, and FISH. Results are then correlated with patient-outcome variables and known risk factors, namely gender, age at diagnosis, tumor location infratentorial vs. supratentorial), tumor grade (differentiated vs anaplastic), and extent of surgery as well as pathologic variables.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies tumor samples from patients with ependymoma treated on the Children Oncology Group ACNS0121 trial. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the prognostic role of histopathological variables, in particular cellular density, mitotic count, and tumor cell invasion in intracranial pediatric ependymomas.

II. To study whether hTERT expression and telomere dysfunction correlate with progression-free survival (PFS) and overall survival (OS) in pediatric intracranial ependymoma.

III. To perform a genome-wide copy number screen and validation of copy number abnormalities (CNAs) on formalin-fixed paraffin-embedded (FFPE) ependymomas using Affymetrix Molecular Inversion Probe (MIP) arrays and interphase fluorescence in situ hybridization (iFISH). IV. To evaluate associations between infiltration of immune markers and PFS as well as OS in pediatric ependymoma.

V. To examine the role of 1q gain and 9p deletion in pediatric ependymomas by exploring their association with PFS and OS in a multivariable model.

VI. To establish the frequency and clinicopathological associations of mutations in genes involved in Notch pathway signaling.

OUTLINE:

Archived tumor tissue samples are analyzed for cellular density, mitotic count, tumor cell invasion, hTERT expression, telomere dysfunction, 1q gain, 9p deletion, and genetic mutations by IHC, Affymetrix Molecular Inversion Probe (MIP) arrays, and fluorescence in situ hybridization (FISH). Results are then correlated with patient-outcome variables and known risk factors, namely gender, age at diagnosis, tumor location infratentorial vs. supratentorial), tumor grade (differentiated vs anaplastic), and extent of surgery as well as pathologic variables.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ependymoma and treated on COG-ACNS0121
* Previously collected tumor samples banked at the Children Oncology Group BioPathology

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with ependymoma treated on the Children Oncology Group ACNS0121 trial
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
PFS | From the time of study enrollment to disease progression, disease relapse or death from any cause
  The multivariable Cox model and cumulative incidence regression models will be used. Associations between the biology markers and outcome variables will be studied in a single-variable setting as well as via multivariable Cox models.
OS | From the time of study enrollment to death from any cause
  The multivariable Cox model and cumulative incidence regression models will be used. Associations between the biology markers and outcome variables will be studied in a single-variable setting as well as via multivariable Cox models.

CONTACTS AND LOCATIONS:
Overall Officials: Uri Tabori, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States